CLINICAL TRIAL: NCT05016102
Title: Different Exercise Types on Inhibitory Control in Children With ADHD
Brief Title: Exercise Enhances Brain Function in Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201404EM038
Record Dates: First submitted 2020-10-09; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Exercise; ADHD; Executive Dysfunction
Keywords: intensity; exercise; executive function; ADHD
MeSH Terms: conditions — Motor Activity; Attention Deficit Disorder with Hyperactivity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control condition (Other): 30 min to watching exercise-related video
  Interventions: Other: Exercise type
- Aerobic exercise condition (Other): 20 minutes of moderate-intensity exercise on treadmill
  Interventions: Other: Exercise type
- Resistance exercise condition (Other): One set of 15 repetition 9 muscle exercises dumbbell squat with chair, dumbbell right/left foot lunge, sit-up, push-up, back muscle with superman, dumbbell right/left bicep curl, dumbbell calf raise.
  Interventions: Other: Exercise type

INTERVENTIONS:
Other: Exercise type — Aerobic exercise and Resistance exercise

SUMMARY:
The aim of the study was to investigate the different effects of exercise types on inhibitory control in children with attention-deficit/ hyperactivity disorder.

DETAILED DESCRIPTION:
Study inclusion criteria were as follows: (1) age between 8 and 12 years; (2) diagnosed with ADHD by a pediatric psychiatrist; and (3) no history of brain injury or neurological conditions, such as exhibited epileptic seizures, serious head injuries, and periods of unconsciousness.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 7 and 12 years
2. diagnosed by a pediatric psychiatrist
3. no history of brain injury
4. no neurological conditions

Exclusion Criteria:

1. less than 50% accuracy
2. failed to complete the task
3. cannot follow the instruction

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2013-08-23 (Actual); Primary Completion 2014-03-15 (Actual); Study Completion 2014-03-15 (Actual)

PRIMARY OUTCOMES:
Behavioral performance | around 10-30 minutes after exercise intervention
  reaction time of stroop and simon task following congruent and incongruent condition.

SECONDARY OUTCOMES:
P3 component | around 10-30 minutes after exercise intervention
  P3 of event-related potentials component, a larger P3 amplitude and shorter P3 latency means better performance

OTHER OUTCOMES:
EEG | around 10-30 minutes after exercise intervention
  Alpha power/ event-related desynchronization (ERD)

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Min Hung, Study Chair — Department of Physical Education, National Taiwan Normal University